CLINICAL TRIAL: NCT06000241
Title: Comparison of Same Morning vs Previous Evening Dosing Regimen for Assessment of Quality of Bowel Preparation Under Anesthesia
Brief Title: Comparison of Same Morning vs Previous Evening Dosing Regimen for Assessment of Quality of Bowel Preparation for Colonoscopy Under Anesthesia
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: JS-3388
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-03

CONDITIONS: Bowel Preparation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
220 patients are allocated randomly to the morning group (am group) or the afternoon group (pm group) and assessed by quality of bowel preparation and residual volume gastric residue.

ELIGIBILITY:
Inclusion Criteria:

Patients are able to follow the instructions of bowel preparation and have good ability of walking at least an hour.

Exclusion Criteria:

Clinical diagnosis of obstruction of bowel and sever renal and heart disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants have a cluster of elective EGD and colonoscopy under anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
ottawa score | a day
  Two nurses observe cleaning of three parts of colon and give a score for each.
gastric residual volume | 30 minutes
  Gastric contents are suctioned and measured.
colonic residual volume | 30 minutes
  Colonic fluids are suctioned and measured.

SECONDARY OUTCOMES:
reflux | 60mins
  incidence of reflux during both the EGD and colonoscopy
adenoma detection rate | a day
  percentages of patients screened with colonic adenoma in total patients

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Peking Union Medical Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing